CLINICAL TRIAL: NCT01314664
Title: A PROSPECTIVE REGISTRY TO ASSESS THE EFFECTIVENESS AND LOCAL TOLERABILITY OF INTRAVESICAL VALRUBICIN IN SUBJECTS WITH NON-MUSCLE INVASIVE BLADDER CANCER (NMIBC)
Status: Terminated | Type: Observational
Why Stopped: Business decision, not safety related
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: EN3329-402
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Bladder Cancer; CIS
Keywords: Non-Muscle Invasive Bladder Cancer; CIS; BCG Refractory
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to observe and describe the effectiveness and local tolerability of intravesical treatment with valrubicin for non-muscle invasive bladder cancer (NMIBC) in a cohort of subjects treated under routine practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years of age and older
* Diagnosed with NMIBC
* Prescribed intravesical valrubicin to treat NMIBC
* Understood and signed Informed Consent to participate

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects who will be receiving intravesical valrubicin treatment for NMIBC
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Kirby, PhD, Study Director — Endo
Locations (11):
- United States (11):
  - BCG Oncology, Phoenix, Arizona
  - Urology Research Network, Hialeah, Florida
  - Advanced Urology Association of Florida, Vero Beach, Florida
  - Kansas City Urology Care, Overland Park, Kansas
  - Delaware Valley Urology, Sewell, New Jersey
  - Delaware Valley Urology, Voorhees Township, New Jersey
  - Long Island Urological Associates, Bethpage, New York
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology Associates of North Texas, Arlington, Texas
  - Urology Clinics of North Texas, Dallas, Texas